CLINICAL TRIAL: NCT04455282
Title: CIRCULATing Biomarkers for Individualized Surgical Therapy in gastroEsophageal Cancer - Phase 1
Acronym: CIRCULATE1
Status: Recruiting | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: University Hospital of Cologne (Other)
Responsible Party: Principal Investigator, Univ.-Prof. Dr. med. Nikolas H. Stoecklein, Head of Experimental Surgical Oncology, Heinrich-Heine University, Duesseldorf
Other Study IDs: 2020-06-BS
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Cancer of Esophagus; Esophagogastric Junction Disorder
Keywords: Circulating Biomarkers; CTC; tdEVs; ctDNA
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, tumor material
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an exploratory observational biomarker study in approximately 100 eligible patients with resectable adenocarcinomas of the esophagus and gastro- esophageal junction (GEJ) type I-II (GEAC) to investigate the difference deletion frequency of circulating tumor cells (CTCs) between peripheral veins and tumor-draining veins (primary endpoint), prognostic value, relevance of a set of two additional blood-based biomarkers analyzed from a single blood sampling tube (secondary endpoints). The underlying hypothesis is that the biomarker alone or in combination improve preoperative staging and help to identify patients at risk for metastasis. This should enable a better stratification of GEAC patients to neo-adjuvant treatment, (intensified) peri-operative treatment, or even surgery alone, in selected cases. The data of the CIRCULATE study shall be used design subsequent studies testing the predictive role of these biomarkers for surgical management. Patients will provide blood samples and lymphatic fluid during the operation and annual blood samples during clinical follow up of 5 years.

DETAILED DESCRIPTION:
This is an exploratory observational biomarker study. Around 20 mL of blood will be collected from a peripheral vein and additional 40 mL from tumor draining veins. In addition, around 5 mL of lymphatic fluid will be collected from the thoracic duct, when exposed and opened during the surgical resection. Annual blood draws (20 mL) will be performed during routine clinical follow-up or at the time point when the patients develops a (metastatic) relapse. A one tube protocol will be performed from each blood sample to assess CTCs and tumor derived extracellular Vesicles (tdEVs) using CELLSEARCH® and ACCEPT (https://github.com/LeonieZ/ACCEPT/blob/master/ACCEPT.m). In addition, tumor cells will be enumerated by CELLSEARCH® in the lymphatic fluid. ctDNA will be extracted from plasma of each blood collection tube and analyzed by mFAST-SeqS. If the mutational status of the primary tumor is known, deep sequencing of ctDNA will be applied for mutation tracking at a later time point. Tissue resected during the surgical procedure and not required for routine pathology will be collected into a biobank (cry-conserved and formalin fixed and paraffin embedded (FFPE).

ELIGIBILITY:
Inclusion Criteria:

* histologically proven adenocarcinoma of the GEJ type I and II, resectable, non-metastatic tumor
* age ≥18
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2,
* American Society of Anesthesiologists (ASA) < 4.
* pre-treatment stage cT1N+ M0 or cT2-4a N0/N+, M0 GEJ type I and II adenocarcinomas can be included. In case of stage cT4a, curative resectability has to be explicitly verified by the local surgical investigator prior inclusion.
* Written informed consent and the ability to understand the nature of the study and the study-related procedures and to comply with them has to be ensured.

Exclusion Criteria:

* tumors of squamous, adenosquamous or other non-adenocarcinoma histology
* patients with inoperable or metastatic GEJ type I and II adenocarcinoma, GEJ type I and II adenocarcinoma staged cT1N0 and cT4b, GEJ type I and II cT4a evaluated as not curatively resectable by the local surgical investigator
* unsigned informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The targeted study population of CIRCULATE1 are 100 patients (see 2.3) with resectable GEAC (GEJ type I-II) undergoing surgery with curative intention. The patients will be recruited and screened consecutively by trained surgeons involved into the CIRCULATE study. Patients are recruited to participate in this study at the outpatient clinic
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Difference in CTC detection rate between peripheral and tumor draining veins. | 24 months
  The difference between the CTC positivity rate (≥1 CTC / 7.5 mL) in blood samples of tumor-draining veins compared to the CTC positivity rate in peripheral blood. The positivity fraction and CTC number per 7.5 mL in tumor draining veins and peripheral blood samples will be determined by CellSearch.

SECONDARY OUTCOMES:
tdEVs | 24 months
  1. The tdEV number per 7.5 mL determined from CellSearch images using the ACCEPT software tool and the fraction of tdEVs positive patients (a cut-off threshold will be applied)(de Wit, 2019). 2. The difference between tdEV measurement in the tumor-draining veins and the peripheral blood will be assessed.
ctDNA | 24 months
  1. The tumor allele frequency measured by the genome-wide mFAST-SeqS assay (Belic, 2015) and the fraction of patients with high tumor allele frequency will be determined. For this, a threshold of 10% tumour allele frequency will be applied to discriminate high allele frequency (>10%) from low allele frequency (≤10%) cases (Belic, 2015; de Wit, 2019). 2. The difference between ctDNA measurement in the tumor-draining veins and the peripheral blood will be assessed.
Clinical correlation | 84 months
  Correlation of any of the biomarker or in combination with clinical parameters and with patient clinical outcome (OS and RFS)
Dynamic Biobank | 24 months
  The number of tumor tissues (primary tumor, lymph node metastasis, biopsy material), isolated CELLSEARCH® CTCs and plasma/ctDNA samples generated from CIRCULATE1 and stored in the respective biobanks from the University Hospital of Cologne and from University Hospital Düsseldorf.

CONTACTS AND LOCATIONS:
Overall Officials: Nikolas Stoecklein, MD, Principal Investigator — Surgery, University Hospital Düsseldorf Germany; Christiane Bruns, MD, Principal Investigator — Surgery, University Hospital Cologne
Locations (2):
- Germany (2):
  - University Hospital Cologne, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Münster, Münster, North-Rhine Westfalia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] de Wit S, Rossi E, Weber S, Tamminga M, Manicone M, Swennenhuis JF, Groothuis-Oudshoorn CGM, Vidotto R, Facchinetti A, Zeune LL, Schuuring E, Zamarchi R, Hiltermann TJN, Speicher MR, Heitzer E, Terstappen LWMM, Groen HJM. Single tube liquid biopsy for advanced non-small cell lung cancer. Int J Cancer. 2019 Jun 15;144(12):3127-3137. doi: 10.1002/ijc.32056. Epub 2019 Jan 28. PMID 30536653
- [Background] Belic J, Koch M, Ulz P, Auer M, Gerhalter T, Mohan S, Fischereder K, Petru E, Bauernhofer T, Geigl JB, Speicher MR, Heitzer E. Rapid Identification of Plasma DNA Samples with Increased ctDNA Levels by a Modified FAST-SeqS Approach. Clin Chem. 2015 Jun;61(6):838-49. doi: 10.1373/clinchem.2014.234286. Epub 2015 Apr 20. PMID 25896989
- [Background] Reeh M, Effenberger KE, Koenig AM, Riethdorf S, Eichstadt D, Vettorazzi E, Uzunoglu FG, Vashist YK, Izbicki JR, Pantel K, Bockhorn M. Circulating Tumor Cells as a Biomarker for Preoperative Prognostic Staging in Patients With Esophageal Cancer. Ann Surg. 2015 Jun;261(6):1124-30. doi: 10.1097/SLA.0000000000001130. PMID 25607767
- [Background] Pernot S, Badoual C, Terme M, Castan F, Cazes A, Bouche O, Bennouna J, Francois E, Ghiringhelli F, De La Fouchardiere C, Samalin E, Bachet JB, Borg C, Ducreux M, Marcheteau E, Stanbury T, Gourgou S, Malka D, Taieb J. Dynamic evaluation of circulating tumour cells in patients with advanced gastric and oesogastric junction adenocarcinoma: Prognostic value and early assessment of therapeutic effects. Eur J Cancer. 2017 Jul;79:15-22. doi: 10.1016/j.ejca.2017.03.036. Epub 2017 Apr 26. PMID 28456090
- [Background] Buscail E, Chiche L, Laurent C, Vendrely V, Denost Q, Denis J, Thumerel M, Lacorte JM, Bedel A, Moreau-Gaudry F, Dabernat S, Alix-Panabieres C. Tumor-proximal liquid biopsy to improve diagnostic and prognostic performances of circulating tumor cells. Mol Oncol. 2019 Sep;13(9):1811-1826. doi: 10.1002/1878-0261.12534. Epub 2019 Jul 25. PMID 31216108